CLINICAL TRIAL: NCT04442230
Title: Phase 2, Double-blind, Randomized, Placebo-controlled Study of NasoVAX in the Prevention of Clinical Worsening in Patients With Early Coronavirus Infectious Disease 2019 (COVID-19)
Brief Title: NasoVAX in Patients With Early Coronavirus Infectious Disease 2019 (COVID-19)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment
Sponsor: Altimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALT-601-201
Record Dates: First submitted 2020-06-17; First posted 2020-06-22 (Actual); Results first posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-02

CONDITIONS: Coronavirus Infection
Keywords: COVID-19; SARS-CoV-2
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NasoVAX (Experimental): Participants will receive a single intranasal dose of NasoVAX on Day 1 (enrollment).
  Interventions: Biological: NasoVAX
- Placebo (Placebo Comparator): Participants will receive a single intranasal dose of placebo on Day 1 (enrollment).
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: NasoVAX — NasoVAX consists of replication-deficient adenovirus vectors in suspension
  Arms: NasoVAX
Other: Placebo — Normal saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of NasoVAX in preventing worsening of symptoms and hospitalization in patients with early COVID-19.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patient volunteers that have given written informed consent will undergo screening to determine eligibility for study entry. If the patient qualifies for the study, they will be randomized in a double-blind manner in a 1:1 ratio to receive NasoVAX or placebo. On the same day of qualifying into the study, the patient will be administered the investigational drug (either NasoVAX or placebo).

The patient will return home for the remainder of the study. During this period, the patient will be monitored remotely by the study center for clinical status. The patient will also be contacted by study center personnel by telephone to ask about use of any medications and changes in health including information about any hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide informed consent (Patients themselves must provide written informed consent before the performance of any study-related procedures, and surrogate consent by family members, designated legal representatives or caregivers will not be permitted).
2. Men and women 18 years of age and older
3. Early COVID-19, defined as one or more symptom(s) of fever (oral temperature ≥ 100.4 degrees F), cough, or shortness of breath, onset of these symptoms within 72 hours of screening, and confirmation of SARS-CoV-2 infection by a polymerase chain reaction (PCR)-based or rapid antigen diagnostic.
4. Resting SpO2 ≥ 96.0% on room air on two successive measurements
5. For women of childbearing potential (women who are not permanently sterile [documented hysterectomy, bilateral tubal ligation, salpingectomy, or oophorectomy] or postmenopausal [12 months with no menses without an alternative medical cause])

   * Negative urine pregnancy test at Screening
   * Willingness to practice a highly effective method of contraception that includes, but is not limited to, abstinence, sex only with persons of the same sex, monogamous relationship with a postmenopausal partner, monogamous relationship with vasectomized partner, vasectomy, licensed hormonal methods, intrauterine device, or consistent use of a barrier method (eg, condom, diaphragm) with spermicide for 28 days after the last dose of study drug
6. For men with sexual partners of childbearing potential, willingness to practice a highly effective method of contraception, as defined above, for 45 days after the last dose of study drug
7. Ability and willingness to comply with all aspects of the study, including reliable internet access, through the entire study period

Exclusion Criteria:

1. Pregnant or lactating women or planning to conceive a child during the next 3 months
2. Resting respiratory rate >20 breaths/min on room air or resting pulse rate ≥ 125 beats per minute
3. A rapidly worsening course that in the opinion of the Investigator or treating medical practitioner would lead to hospitalization within the next 24-48 hours
4. Any chronic pulmonary disease, including chronic obstructive pulmonary disease and asthma, or other respiratory diseases that could exacerbate independent of COVID-19
5. The following risk factors for severe COVID-19 (Cohorts 1 and 2 only) (Centers for Disease Control 2020), which based on ongoing review of efficacy and safety data, the DMC may remove part or all of these risk factors if preliminary data show no signal for adverse or paradoxical effects:

   1. Severe obesity, defined as body mass index ≥ 40 kg/m2
   2. History of:

      * Severe cardiovascular disease, including but not limited to congestive heart failure, coronary artery disease, congenital heart disease, cardiomyopathies, or pulmonary hypertension
      * Diabetes mellitus
      * Chronic or current vaping or cigarette smoking
      * Chronic kidney disease requiring dialysis
      * Chronic liver disease, including but not limited to chronic viral hepatitis, non-alcoholic steatohepatitis, or cirrhosis of any cause
      * Hemoglobin disorder, including sickle cell disease and thalassemia
6. History of Bell's Palsy
7. Nasal conditions that might affect the suitability of intranasal medication, such as a history of chronic rhinitis, nasal septal defect, cleft palate, nasal polyps, or nasal surgery other than cosmetic rhinoplasty.
8. Use of hydroxychloroquine within the past 4 months, chloroquine with the past 9 months, or other investigational agents for COVID-19 within the past 30 days
9. History of conditions associated with immunocompromise, including but not limited to poorly controlled HIV, or treatments known to affect the immune system, including but not limited to oral or intravenous corticosteroids, alkylating drugs, antimetabolites, cytotoxic drugs, radiation, immune-modulating biologics (including interleukin [IL]-6, IL-12, Janus kinase inhibitors or antagonists), and cancer treatments, within 30 days of Screening, or anticipated use within 6 months following participation in this study
10. Any medical, psychiatric, or social condition or occupational or other responsibility that in the judgment of the Investigator would interfere with or serve as a contraindication to protocol adherence, assessment of safety (including reactogenicity), or a patient's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Miami Dade Medical Research Institute, Miami, Florida
  - Infinite Clinical Trials, Morrow, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - Carolina Institute for Clinical Research, Fayetteville, North Carolina
  - Next Level Urgent Care, Houston, Texas
  - Centex Studies, Houston, Texas
  - Centex Studies, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NasoVAX | Placebo
Started | 23 | 25
Completed | 23 | 24
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | NasoVAX | Placebo | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (14.05) | 42.6 (14.98) | 42.2 (14.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 14 | 16 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 22 | 43
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 23 | 24 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 25 | 48
Risk factors for severe COVID-19 [Count of Participants; unit: Participants]
  Risk factors present | 2 | 1 | 3
  No risk factors present | 21 | 24 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Clinical Worsening
Description: Absolute 4.0% decrease from baseline in resting SpO2 on two consecutive measurements
Time Frame: Day 1 to Day 14
Population: Modified intent-to-treat population (all randomized patients who received any amount of study drug and had a Baseline and at least one post-baseline resting SpO2 measurement)
Measure: Count of Participants; unit: Participants
Arm/Group | NasoVAX | Placebo
Number analyzed (Participants) | 23 | 25
Participants | 3 | 2
Statistical Analysis 1: Comparison: NasoVAX vs Placebo; The p-values from significance tests were obtained at a one-sided significance level of 0.025; Test type: Superiority; p = 0.6602, Fisher Exact

2. Secondary Outcome: Maximal Severity of COVID-19 After Treatment
Description: Percentage of patients requiring hospitalization
Time Frame: Day 1 to Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | NasoVAX | Placebo
Number analyzed (Participants) | 23 | 25
Participants | 0 | 0

3. Secondary Outcome: All-cause Mortality
Description: All-cause mortality through Day 42
Time Frame: Day 1 to Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | NasoVAX | Placebo
Number analyzed (Participants) | 23 | 25
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days, or up to 42 days for subject hospitalized for COVID-19 at Day 28
Arm/Group | NasoVAX | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 22/23 | 18/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NasoVAX (N=23) | Placebo (N=25)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 5 (7)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 6 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 8 (10) | 2 (2)
Fatigue (Gastrointestinal disorders) | 4 (4) | 3 (4)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 8 (9)
Nausea (Gastrointestinal disorders) | 5 (7) | 5 (5)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1)
Anosmia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All information provided regarding the study, as well as all information collected/documented during the course of the study, will be regarded as confidential. The Investigator agrees not to disclose such information in any way without prior written permission from the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/30/NCT04442230/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT04442230/SAP_001.pdf